CLINICAL TRIAL: NCT05380583
Title: Treatment Engagement in Families With Substance Use and Psychosis: A Pilot Study
Brief Title: Community Reinforcement and Family Training for Early Psychosis (CRAFT-EP) and Substance Use: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Julie McCarthy, Ph.D., Assistant Professor of Psychology, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020P000220-A; K23DA050808 (NIH)
Record Dates: First submitted 2022-05-09; First posted 2022-05-19 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Psychosis; Substance Use; Substance Use Disorders; Family; Cannabis; Marijuana; Alcohol; Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Mental Disorder
MeSH Terms: conditions — Psychotic Disorders; Substance-Related Disorders; Marijuana Abuse; Schizophrenia; Bipolar Disorder; Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRAFT-EP + TAU (Experimental): Community Reinforcement and Family Training for Early Psychosis (CRAFT-EP) with 8 weekly sessions of 60-90-minute coaching + Treatment as Usual (TAU).
  Interventions: Behavioral: CRAFT-EP; Behavioral: TAU
- Treatment as Usual (Active Comparator): Treatment as Usual
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: CRAFT-EP — CRAFT-EP is a behavioral intervention delivered via telehealth with the option for one in-person session (when local guidelines allow in-person care without masks). The coaching session topics include self-care, communication, functional analysis, positive reinforcement, treatment engagement, natural consequences, problem solving, and planning next steps. The intervention is designed for families of individuals experiencing psychosis and substance use who are enrolled or seeking enrollment in early psychosis outpatient services. Participants will be asked to complete assessments at pre-, mid- (approximately week 4), post-intervention, and a follow-up assessment approximately 12 weeks post-intervention.
  Other Names: Community Reinforcement and Family Training for Early Psychosis (CRAFT-EP)
  Arms: CRAFT-EP + TAU
Behavioral: TAU — Participants may continue to receive their ongoing treatment, if any, which may include psychosocial and/or pharmacological interventions.
  Other Names: Treatment as Usual (TAU)

SUMMARY:
The purpose of this study is to evaluate Community Reinforcement and Family Training for Early Psychosis (CRAFT-EP) for families experiencing early psychosis and substance use delivered exclusively or primarily via telehealth (video conferencing).

DETAILED DESCRIPTION:
The intervention aims to improve treatment engagement, substance use patterns, and family wellbeing. To assess preliminary outcomes of the intervention, this study compares CRAFT-EP plus treatment as usual (TAU) compared to TAU alone. Family members will be randomized to CRAFT-EP + TAU or TAU alone. Data on family members and clients with psychosis will be collected for assessment purposes; if a client with psychosis does not have a family member participating in the study, the client with psychosis will be automatically be assigned to the TAU alone group. Total target enrollment is 40 family members and 40 clients with psychosis. Given that family members may participate without a corresponding client with psychosis due to fear of disclosing their participation in the study to the client or client lack of interest, and because the intervention works directly with family members and indirectly with clients, data collected from clients with or without a corresponding family member participating in the study will be hypothesis generating.

ELIGIBILITY:
Inclusion Criteria for Family Members:

* Ages 18-70.
* Having a relative who:

  1. Is a client with early course psychosis (schizophrenia, schizoaffective disorder, schizophreniform, psychosis not otherwise specified (NOS), delusional disorder, brief psychotic disorder, major depression with psychosis, and bipolar disorder with psychosis (as reported by family member, clinician, or chart review)) with first onset in the past 6 years, and
  2. Used alcohol or cannabis in the past 30 days and/or has no apparent immediate interest in abstinence (responding "No" to "Do you think they want to quit right now?" in reference to overall substance use).
  3. Family member has concerns about the relative's substance use.
* The person(s) who can best describe the client with psychosis.
* At least 4 days per month contact with the client.
* Access to a computer with internet or mobile phone with video conferencing capabilities.
* Ability to provide written informed consent.
* Speak and read English.

Exclusion Criteria for Family Members:

* DSM-5 moderate or severe substance use disorder in the past year.
* Lifetime psychotic disorder.
* History of domestic violence with the client relative that would interfere with the ability to safely follow through with the intervention plan.
* Psychiatric, cognitive, or medical impairments that would interfere with the ability to follow through with the intervention plan.
* Prior participation of a family member of the client in the study program.
* Significant prior experience with CRAFT (e.g., having completed a CRAFT course prior to study enrollment)

Inclusion Criteria for Client Relatives:

* Ages 18-35.
* First episode psychosis onset in the past 6 years with a Diagnostic and Statistical Manual (DSM)-5 diagnosis of affective (bipolar disorder or major depressive disorder with psychotic features) or non- affective psychosis (schizophrenia spectrum disorder)
* Used alcohol or cannabis in the past 30 days and/or has no apparent immediate interest in abstinence (responding "No" to "Do you want to quit right now?" in reference to overall substance use).
* They or others have concerns about the client's substance use.
* Ability to provide written informed consent (or assent with their legal guardian providing informed consent)
* Speak and read English.

Exclusion Criteria for Client Relatives:

- N/A

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Family Wellbeing: Depression | Baseline, mid-intervention (week 4), post-intervention (week 8)
  Beck Depression Inventory-II total; scores range from 0 to 63 with higher scores representing more severe depressive symptoms.

SECONDARY OUTCOMES:
Family Wellbeing: Anxiety | Baseline, mid-intervention (week 4), post-intervention (week 8)
  State-Trait Anxiety Inventory-Short Form; total scores range from 6 to 24 with higher scores representing more severe anxiety symptoms.
Family Wellbeing: Relationship | Baseline, mid-intervention (week 4), post-intervention (week 8)
  General Happiness item on Relationship Happiness Scale; scores range from 1 to 10 with higher scores representing greater relationship happiness.

CONTACTS AND LOCATIONS:
Overall Officials: Julie M McCarthy, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No